CLINICAL TRIAL: NCT03890120
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of Cilofexor in Non-Cirrhotic Subjects With Primary Sclerosing Cholangitis
Brief Title: Study of Cilofexor in Adults With Primary Sclerosing Cholangitis
Acronym: PRIMIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following recommendation of the external Data Monitoring Committee, after it reviewed the results of a planned interim futility analysis.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-428-4194; 2019-000204-14 (EudraCT Number); jRCT2080224728 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — cilofexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cilofexor 100 mg (Blinded Phase) (Experimental): Participants received cilofexor 100 mg tablet, orally, once daily for up to 100.3 weeks.
  Interventions: Drug: Cilofexor
- Placebo (Blinded Phase) (Placebo Comparator): Participants received placebo to match cilofexor 100 mg tablet, orally, once daily for up to 98.1 weeks.
  Interventions: Drug: Placebo
- Cilofexor From Cilofexor 100 mg (OLE Phase) (Experimental): Participants who received cilofexor in blinded phase and had entered the open-label extension (OLE) phase received open-label cilofexor 100 mg tablet, orally, once daily for up to 44.7 weeks.
  Interventions: Drug: Cilofexor
- Cilofexor From Placebo (OLE Phase) (Experimental): Participants who received placebo in blinded phase and had entered the OLE phase received open-label cilofexor 100 mg tablet, orally, once daily for up to 45.0 weeks.
  Interventions: Drug: Cilofexor

INTERVENTIONS:
Drug: Cilofexor — 100 mg tablet administered orally once daily
  Other Names: GS-9674
  Arms: Cilofexor 100 mg (Blinded Phase); Cilofexor From Cilofexor 100 mg (OLE Phase); Cilofexor From Placebo (OLE Phase)
Drug: Placebo — Tablet administered orally once daily
  Arms: Placebo (Blinded Phase)

SUMMARY:
The primary objective of this study is to evaluate whether cilofexor reduces the risk of fibrosis progression among non-cirrhotic adults with primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of large duct PSC
* Liver biopsy at screening that is deemed acceptable for interpretation and demonstrates stage F0 - F3 fibrosis in the opinion of the central reader
* Individual has the following laboratory parameters at the screening visit, as determined by the central laboratory:

  * Platelet count ≥ 150,000/mm^3
  * Estimated glomerular filtration rate (eGFR) ≥ 30 milliliter/minute (mL/min), as calculated by the Cockcroft-Gault equation
  * Alanine transaminase (ALT) ≤ 8 x upper limit of the normal range (ULN)
  * Total bilirubin < 2 mg/dL, unless the individual is known to have Gilbert's syndrome or hemolytic anemia
  * International normalized ratio (INR) ≤ 1.4, unless due to therapeutic anticoagulation
  * Negative anti-mitochondrial antibody

Key Exclusion Criteria:

* Current or prior history of any of the following:

  * Cirrhosis
  * Liver transplantation
  * Cholangiocarcinoma or hepatocellular carcinoma (HCC)
  * Ascending cholangitis within 30 days of screening
* Presence of a percutaneous drain or biliary stent
* Other causes of liver disease
* Current or prior history of unstable cardiovascular disease
* Current moderate to severe inflammatory bowel disease (IBD) (including ulcerative colitis, Crohn's disease, and indeterminate colitis)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (201):
- United States (82):
  - Institute For Liver Health, Glendale, Arizona
  - The Institute for Liver Heath, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - Altman Clinical and Translational Research Institute (Clinic), La Jolla, California
  - Scripps Clinic/Green Hospital, La Jolla, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Stanford Hospital, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California, Davis Medical Center (study visits), Sacramento, California
  - Sutter Pacific Medical Foundation - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco Liver Clinic, San Francisco, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital; Clinical Research Unit, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center (outpatient clinic), Chicago, Illinois
  - NorthShore University Healthsystem, Evanston, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Gastroenterology, PA, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Saint Louis University, Gastroenterology & Hepatology, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers New Jersey Medical School - Doctors Office Center, Newark, New Jersey
  - Northwell Health Center for Liver Diseases and Transplantation, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Center for Liver Disease and Transplantation, Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - The University of NC at Chapel Hill, Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Carolinas Medical Center - Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Holmes Hospital, Cincinnati, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Annette & Harold C. Simmons Transplant Institute @ Baylor University Medical Center at Dallas, Dallas, Texas
  - Baylor Scott & White Medical Center at Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Spring Gastroenterology Associates, Humble, Texas
  - San Antonio Military Medical Center, Gastro/Hepatology, San Antonio, Texas
  - Intermountain Medical Center - Transplant Services, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Verity Research Inc., Fairfax, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Virginia Commonwealth University Clinical Research Services Unit, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
- Australia (13):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Coral Sea Clinical Research Institute - Mackay, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Landeskrankenanstalten-Betriebsgesellscaft - KABEG, Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Allgemeines Krankenhaus Wien, Vienna
- Belgium (6):
  - Hôpital Erasme - ULB, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège Site Sart Tilman, Liège
- Canada (13):
  - William Osler Health System - Brampton Civic Hospital, Brampton
  - University of Calgary Liver Unit - Heritage Medical Research Clinic (HMRC), Calgary
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre (WMC), Edmonton
  - Queen Elizabeth II Health Sciences Centre, Nova Scotia Health Authority, Halifax
  - St. Joseph's Healthcare Hamilton, Hamilton
  - McMaster University Medical Center, Hamilton
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal
  - Chronic Viral Illness Service/McGill University Health Centre (MUHC), Montreal
  - Toronto General Hospital - Toronto Centre for Liver Disease (TCLD), Toronto
  - Toronto Liver Centre, Toronto
  - Gordon and Leslie Diamond Health Care Centre, Vancouver General Hospital, UBC Division of Gastroenterology, Vancouver
  - (G.I.R.I.) GI Research Institute, Vancouver
  - University of Manitoba/Health Sciences Centre, Winnipeg
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Copenhagen University Hospital - Hvidovre, København Ø
- Finland (2):
  - Helsinki University Hospital, Endoscopy Unit, Gastroenterology Outpatient clinic, Meilahden tomisairaala, Helsinki
  - Turku University Hospital, Gastroenterology Outpatient Clinic, Turku
- France (13):
  - Hôpital Saint-Eloi, Montpellier, Herault
  - CHU Amiens-Picardie Hôpital Sud, Amiens
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, CHRU Lille
  - Hôpital Henri Mondor, Créteil
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Saint-Joseph, Marseille
  - Hopital Saint Antoine, Paris
  - CHU Bordeaux-Hopital Haut-Leveque, Pessac
  - Hopital Robert Debré - Centre Hospitalier Universitaire de Reims, Reims
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU de Toulouse Hopital Ranguiel, Toulouse
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - Hopital Paul Brousse, Villejuif
- Germany (10):
  - GASTRO-Studien GbR, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Medizinische Hochscule Hannover, Hanover
  - Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin II, Gastroenterologie und Hepatologie, Homburg
  - Gastroenterologisch-Hepatologisches Zentrum Kiel, Kiel
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz
  - Universitätsmedizin Mannheim, II. Medizinische Klinik, Mannheim
- Israel (8):
  - Emek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - IRCCS Ospedale Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Dipartimento Gastroenterologico e dei Trapianti, Ancona
  - Azienda Ospedaliero Universitaria di Moderna, Ospedale di Baggiovara, Bologna
  - Ca'Granda Ospedale Maggiore Policlinico UOC Gastroenterologia ed Epatologia, Milan
  - Medicina Interna 1, Novara
  - Azienda Ospedale Universita Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico P. Giaccone, Palermo
  - Azienda Ospedaliero-Universitaria Pisana - Unità Operativa Epatologia, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - U.O.C. Gatroenterologia, Rozzano
  - Istituto Clinico Humanitas - Unita Operativa di Epatologia, Rozzano (Milan)
- Japan (10):
  - Chiba University Hospital, Chiba
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - Okayama University Hospital, Okayama
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai
  - Osaka University Hospital, Suita
  - Juntendo University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Ehime University Hospital, Toon-Shi
  - Yamagata University Hospital, Yamagata
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Universitatsspital Bern, Bern
  - Epatocentro Ticino SA, Lugano
  - Universitatsspital Zurich, Zurich
- United Kingdom (12):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Aintree University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trauner M, Chung C, Sterling K, Liu X, Lu X, Xu J, Tempany-Afdhal C, Goodman ZD, Farkkila M, Tanaka A, Trivedi P, Kowdley KV, Bowlus CL, Levy C, Myers RP. PRIMIS: design of a pivotal, randomized, phase 3 study evaluating the safety and efficacy of the nonsteroidal farnesoid X receptor agonist cilofexor in noncirrhotic patients with primary sclerosing cholangitis. BMC Gastroenterol. 2023 Mar 15;23(1):75. doi: 10.1186/s12876-023-02653-2. PMID 36922785
- [Background] Trauner M, Levy C, Tanaka A, Goodman Z, Thorburn D, et al. A Phase 3 Randomized, Double-blind, Placebo-controlled Study Evaluation the Efficacy and Safety of Cilofexor in Patients With Non-cirrhotic Patients With Primary Sclerosing Cholangitis. J Hepatol. 2023 June;78(S1):S12-S13.
- [Derived] Trauner M, Levy C, Tanaka A, Goodman Z, Thorburn D, Joshi D, Salminen K, Yimam K, Isayama H, Montano-Loza AJ, Caldwell S, Danta M, Farkkila M, Gallegos-Orozco JF, Gordon SC, Hinrichsen H, Invernizzi P, Vuppalanchi R, Zhu K, Xu J, Liu X, Lu X, Crans G, Bolbolan S, Boyette L, Alani M, Barchuk WT, Watkins TR, Genovese MC, Bowlus CL. Cilofexor in non-cirrhotic primary sclerosing cholangitis (PRIMIS): a randomised, double-blind, multicentre, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2026 Jan;11(1):46-58. doi: 10.1016/S2468-1253(25)00208-0. Epub 2025 Oct 28. PMID 41173015
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03890120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, North America, Oceania, and Asia.
Pre-assignment Details: 587 participants were screened.
Period: Blinded Treatment Phase (100.3 Weeks)
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase) | Cilofexor From Cilofexor 100 mg (OLE Phase) | Cilofexor From Placebo (OLE Phase)
Started | 278 | 141 | 0 | 0
Completed | 123 | 66 | 0 | 0
Not Completed | 155 | 75 | 0 | 0
Not completed — Study terminated by sponsor | 119 | 57 | 0 | 0
Not completed — Adverse Event | 17 | 7 | 0 | 0
Not completed — Withdrew consent | 12 | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0 | 0
Not completed — Investigator's discretion | 1 | 2 | 0 | 0
Not completed — Randomized but never treated | 1 | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Period: Open-Label Extension Phase (45 Weeks)
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase) | Cilofexor From Cilofexor 100 mg (OLE Phase) | Cilofexor From Placebo (OLE Phase)
Started | 0 (Participants who consented to enter the OLE Phase and completed the Blinded Study Phase Week 96 with an evaluable biopsy (noncirrhotic F0, F1, F2, and F3) as determined by the central reader and Blinded Study Phase follow-up visit entered OLE Phase.) | 0 (Participants who consented to enter the OLE Phase and completed the Blinded Study Phase Week 96 with an evaluable biopsy (noncirrhotic F0, F1, F2, and F3) as determined by the central reader and Blinded Study Phase follow-up visit entered OLE Phase.) | 80 (Participants who consented to enter the OLE Phase and completed the Blinded Study Phase Week 96 with an evaluable biopsy (noncirrhotic F0, F1, F2, and F3) as determined by the central reader and Blinded Study Phase follow-up visit entered OLE Phase.) | 45 (Participants who consented to enter the OLE Phase and completed the Blinded Study Phase Week 96 with an evaluable biopsy (noncirrhotic F0, F1, F2, and F3) as determined by the central reader and Blinded Study Phase follow-up visit entered OLE Phase.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 80 | 45
Not completed — Study terminated by sponsor | 0 | 0 | 76 | 42
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrew consent | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase) | Total
Number analyzed (Participants) | 277 | 139 | 416
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 258 | 133 | 391
  >=65 years | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13.1) | 44 (12.8) | 44 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 52 | 159
  Male | 170 | 87 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 258 | 130 | 388
  Unknown or Not Reported | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 228 | 117 | 345
  Race: Asian | 28 | 10 | 38
  Race: Black or African American | 10 | 7 | 17
  Race: Unknown or Not Reported | 6 | 5 | 11
  Race: Other or More Than One Race | 5 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 57 | 171
  Japan | 19 | 8 | 27
  United Kingdom | 11 | 8 | 19
  Switzerland | 2 | 4 | 6
  Spain | 13 | 3 | 16
  New Zealand | 4 | 2 | 6
  Canada | 28 | 10 | 38
  Austria | 3 | 1 | 4
  Belgium | 4 | 2 | 6
  Finland | 11 | 8 | 19
  Denmark | 4 | 3 | 7
  Italy | 17 | 6 | 23
  Israel | 8 | 3 | 11
  Australia | 18 | 13 | 31
  France | 8 | 6 | 14
  Germany | 13 | 5 | 18
Alkaline Phosphatase (ALP) [Mean (Standard Deviation); unit: units per liter (U/L)] | 223 (177.7) | 243 (189.5) | 230 (181.7)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] | 49 (34.1) | 51 (34.6) | 50 (34.2)
Fasting Total Bile Acids [Mean (Standard Deviation); unit: micromoles per liter (μmol/L)] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  micromoles per liter (μmol/L)
    number analyzed (Participants) | 262 | 132 | 394
    (all) | 24.2 (37.57) | 18.6 (22.49) | 22.4 (33.36)
Enhanced Liver Fibrosis (ELF™) Test Score [Mean (Standard Deviation); unit: score on a scale] — The Enhanced Liver Fibrosis (ELF™) test is a composite of three serum biomarkers of hepatobiliary fibrosis: hyaluronic acid, procollagen III amino-terminal peptide, and tissue inhibitor of metalloproteinase. A typical range for ELF™ test scores in PSC is between 6 and 14. Higher ELF™ test scores are associated with more severe liver disease. Population: Participants in the Safety Analysis Set with available data were analyzed.
  score on a scale
    number analyzed (Participants) | 276 | 137 | 413
    (all) | 9.14 (0.910) | 9.13 (0.963) | 9.13 (0.927)
Fibroscan Score [Mean (Standard Deviation); unit: kilopascals (kPa)] — Change in liver stiffness was measured by FibroScan® scores. FibroScan measures liver scarring by measuring the stiffness of the liver. It's normally between 2 and 6 kPa. Many people with liver disease(s) have a result that's higher than the normal range. Higher scores indicate increased scarring of the liver. Population: Participants in the safety analysis set with available data were analyzed.
  kilopascals (kPa)
    number analyzed (Participants) | 253 | 125 | 378
    (all) | 7.8 (4.91) | 8.0 (4.07) | 7.8 (4.64)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression of Liver Fibrosis at Blinded Phase Week 96
Description: Progression of liver fibrosis was defined as having a ≥ 1-stage increase from baseline in fibrosis according to the Ludwig classification at Blinded Phase Week 96. The stages of fibrosis was assessed according to Ludwig classification. Ludwig classification fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=no fibrosis, 4=cirrhosis).
Time Frame: Blinded Phase Week 96
Population: Full Analysis Set included all randomized participants who took at least 1 dose of study drug. Participants in the Full Analysis Set who had nonmissing data at both baseline and Week 96 in the Blinded Study Phase were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 133 | 64
percentage of participants | 30.8 | 32.8
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.4186, Mantel Haenszel; Difference in Percentages = -1.4, 95% CI 2-sided [-15.2 to 12.3] — The difference of cilofexor and placebo,95% confidence interval(CI),and P value(1-sided)were obtained by the stratum-adjusted Mantel-Haenszel (MH) method,with baseline ursodeoxycholic acid(UDCA)use and Ludwig fibrosis stage as stratification factors

2. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) in The Blinded Phase
Description: An AE was any untoward medical occurrence in a clinical study participant administered a study drug that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not the AE is considered related to the study drug. For Blinded Study Phase and OLE Phase, TEAEs were defined as 1 or both of the following: Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date in the Blinded Phase up to 100.3 weeks plus 30 days
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 277 | 139
percentage of participants | 97.1 | 95.0

3. Secondary Outcome: Percentage of Participants Who Experienced TEAEs in The OLE Phase
Description: as for outcome 2
Time Frame: First dose date in the OLE Phase up to 45 weeks plus 30 days
Population: OLE Analysis Set included all participants who took at least 1 dose of study drug in the OLE Phase.
Measure: Number; unit: percentage of participants
Groups:
- Cilofexor From Cilofexor 100 mg (OLE Phase): Participants who received cilofexor in blinded phase and had entered the OLE phase received open-label cilofexor 100 mg tablet, orally, once daily for up to 44.7 weeks.
Arm/Group | Cilofexor From Cilofexor 100 mg (OLE Phase) | Cilofexor From Placebo (OLE Phase)
Number analyzed (Participants) | 80 | 45
percentage of participants | 66.3 | 73.3

4. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Serious Adverse Events (SAEs) in the Blinded Phase
Description: An SAE was defined as an event that, at any dose, results in the following: death, a life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect or a medically important event or reaction.
Time Frame: First dose date in the Blinded Phase up to 100.3 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 277 | 139
percentage of participants | 19.1 | 18.7

5. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent SAEs in the OLE Phase
Description: as for outcome 4
Time Frame: First dose date in the OLE Phase up to 45 weeks plus 30 days
Population: Participants in the OLE Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor From Cilofexor 100 mg (OLE Phase) | Cilofexor From Placebo (OLE Phase)
Number analyzed (Participants) | 80 | 45
percentage of participants | 11.3 | 2.2

6. Secondary Outcome: Change From Baseline in Serum Concentrations of Alkaline Phosphatase (ALP) at Blinded Phase Week 96
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: units per liter (U/L)
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 146 | 74
units per liter (U/L) | 0 [-17 to 16] | 3 [-19 to 25]
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.3884, ANCOVA; Difference in Least Squares Mean (LSM) = -4, 95% CI 2-sided [-28 to 21] — The LSM,95% CI and P-value(1-sided) were obtained by an analysis of covariance(ANCOVA)model with change at Week 96 as dependent variable,baseline value of outcome measure,baseline UDCA use, and baseline Ludwig fibrosis stage as independent variables

7. Secondary Outcome: Change From Baseline in Serum Concentrations of Alanine Aminotransferase (ALT) at Blinded Phase Week 96
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 145 | 74
U/L | -13 [-20 to -6] | -3 [-12 to 6]
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.0390, ANCOVA; Difference in LSM = -9, 95% CI 2-sided [-20 to 1] — The LSM, 95% CI and P-value (1-sided) were obtained by ANCOVA model to evaluate change at Week 96 as the dependent variable, baseline value of the outcome measure, baseline UDCA use, and baseline Ludwig fibrosis stage as independent variables

8. Secondary Outcome: Change From Baseline in Serum Concentrations of Fasting Total Bile Acids at Blinded Phase Week 96
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: micromoles per liter (μmol/L)
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 147 | 74
micromoles per liter (μmol/L) | 7.2 [0.9 to 13.5] | 9.8 [1.8 to 17.9]
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.2845, ANCOVA; Difference in LSM = -2.6, 95% CI 2-sided [-11.6 to 6.4] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Participants With ≥ 25% Relative Reduction in Serum ALP Concentration From Baseline and No Worsening of Fibrosis According to the Ludwig Classification at Blinded Phase Week 96
Description: The stages of fibrosis was assessed according to Ludwig classification. Ludwig classification fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=no fibrosis, 4=cirrhosis).The percentage of participants with ≥ 25% reduction in serum ALP Concentration from baseline and no increase in fibrosis according to the Ludwig Classification at Blinded Phase Week 96 was analyzed.
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data who had nonmissing data at both baseline and Week 96 in the blinded phase were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 122 | 61
percentage of participants | 9.8 | 6.6
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.1978, Mantel Haenszel; Difference in Percentages = 4.1, 95% CI 2-sided [-5.3 to 13.5] — The difference between cilofexor and Placebo, 95% CI, and the p-value (1-sided) were obtained by the stratum-adjusted MH method, with baseline UDCA use and Ludwig fibrosis stage as stratification factors

10. Secondary Outcome: Percentage of Participants With Fibrosis Improvement According to the Ludwig Classification at Blinded Phase Week 96
Description: Fibrosis improvement was defined as having ≥ 1-stage decrease from baseline in fibrosis according to the Ludwig classification score at Blinded Study Phase Week 96. The stages of fibrosis was assessed according to Ludwig classification. Ludwig classification fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=no fibrosis, 4=cirrhosis).
Time Frame: Blinded Phase Week 96
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 133 | 64
percentage of participants | 25.6 | 17.2
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.0797, Mantel Haenszel; Difference in Percentages = 8.9, 95% CI 2-sided [-3.5 to 21.2] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Change From Baseline in Primary Sclerosing Cholangitis (PSC) Symptoms - Module 1 Based on Disease-specific Patient Reported Outcome (PSC-PRO) at Blinded Phase Week 96
Description: The PSC-PRO addressed the severity of common everyday symptoms of PSC (eg, pruritus, fatigue, and right upper quadrant abdominal discomfort); and their functional impact (eg, on physical function, activities of daily living, and work productivity, etc). PSC-PRO module 1 - PSC symptoms contains a total of 12 questions asking about the severity of specific PSC symptoms on a scale of 0 (no symptoms) to 10 (symptoms as bad as you could imagine) with a 24-hour recall period. The total score, which is computed as 12 times the average of nonmissing scores of the 12 questions, can potentially range between 0 and 120, with higher scores indicating more severe symptoms. A positive change from baseline indicates worsening of symptoms.
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 274 | 137
score on a scale
  Baseline | 11 (11.0) | 11 (11.8)
  Change at Blinded Phase Week 96: number analyzed (Participants) | 163 | 78
  Change at Blinded Phase Week 96 | 1 (9.0) | 0 (6.8)
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.7275, ANCOVA; Difference in LSM = 1, 95% CI 2-sided [-1 to 3] — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: Change From Baseline in Enhanced Liver Fibrosis (ELF™ ) Test Score at Blinded Phase Week 96
Description: The Enhanced Liver Fibrosis (ELF™) test is a composite of three serum biomarkers of hepatobiliary fibrosis: hyaluronic acid, procollagen III amino-terminal peptide, and tissue inhibitor of metalloproteinase. A typical range for ELF™ test scores in PSC is between 6 and 14. Higher ELF™ test scores are associated with more severe liver disease. A positive change from baseline indicated worsening of fibrosis.
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 163 | 78
score on a scale | 0.27 [0.16 to 0.38] | 0.30 [0.15 to 0.45]
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.3636, ANCOVA; Difference in LSM = -0.03, 95% CI 2-sided [-0.20 to 0.14] — [estimate comment as in outcome 7, analysis 1]

13. Secondary Outcome: Change From Baseline in Liver Stiffness by FibroScan® at Blinded Phase Week 96
Description: Change in liver stiffness was measured by FibroScan® scores. FibroScan measures liver scarring by measuring the stiffness of the liver. It's normally between 2 and 6 kPa. Many people with liver disease(s) have a result that's higher than the normal range. Higher scores indicate increased scarring of the liver. A positive change from baseline indicates severe liver disease(s).
Time Frame: Baseline, Blinded Phase Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilopascals (kPa)
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase)
Number analyzed (Participants) | 154 | 73
kilopascals (kPa) | 2.4 [1.2 to 3.6] | 2.8 [1.1 to 4.4]
Statistical Analysis 1: Comparison: Cilofexor 100 mg (Blinded Phase) vs Placebo (Blinded Phase); Test type: Superiority; p = 0.3595, ANCOVA; Difference in LSM = -0.3, 95% CI 2-sided [-2.2 to 1.5] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Randomization up to 3.4 years; Adverse events: Blinded Phase: First dose date in the Blinded Phase up to 100.3 weeks plus 30 days; Open-Label Extension (OLE) Phase: First dose date in the OLE Phase up to 45 weeks plus 30 days
Description: All-cause mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse Events: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Cilofexor 100 mg (Blinded Phase) | Placebo (Blinded Phase) | Cilofexor From Cilofexor 100 mg (OLE Phase) | Cilofexor From Placebo (OLE Phase)
All-Cause Mortality (participants affected / at risk) | 2/278 | 0/141 | 0/80 | 0/45
Serious Adverse Events (participants affected / at risk) | 53/277 | 26/139 | 9/80 | 1/45
Other Adverse Events (participants affected / at risk) | 232/277 | 109/139 | 34/80 | 24/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilofexor 100 mg (Blinded Phase) (N=277) | Placebo (Blinded Phase) (N=139) | Cilofexor From Cilofexor 100 mg (OLE Phase) (N=80) | Cilofexor From Placebo (OLE Phase) (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pouchitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 10 | 7 | 2 | 1
Cholangitis acute (Hepatobiliary disorders) | 4 | 0 | 0 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Haemorrhagic cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholangitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 1 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Colorectostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Ligament operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Liver transplant (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilofexor 100 mg (Blinded Phase) (N=277) | Placebo (Blinded Phase) (N=139) | Cilofexor From Cilofexor 100 mg (OLE Phase) (N=80) | Cilofexor From Placebo (OLE Phase) (N=45)
Abdominal distension (Gastrointestinal disorders) | 9 | 9 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 38 | 17 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 40 | 20 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 21 | 11 | 2 | 1
Nausea (Gastrointestinal disorders) | 34 | 16 | 4 | 0
Vomiting (Gastrointestinal disorders) | 12 | 7 | 1 | 0
Fatigue (General disorders) | 34 | 24 | 3 | 0
Pyrexia (General disorders) | 33 | 9 | 3 | 2
Covid-19 (Infections and infestations) | 65 | 26 | 11 | 11
Nasopharyngitis (Infections and infestations) | 15 | 12 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 14 | 7 | 1 | 2
Urinary tract infection (Infections and infestations) | 8 | 5 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 7 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 14 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 8 | 3 | 0
Headache (Nervous system disorders) | 32 | 18 | 1 | 0
Insomnia (Psychiatric disorders) | 14 | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 135 | 50 | 14 | 11
Rash (Skin and subcutaneous tissue disorders) | 16 | 7 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03890120/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT03890120/SAP_001.pdf